CLINICAL TRIAL: NCT05508906
Title: A Phase 1b Open-Label Multicenter Study of OP-1250 (Palazestrant) in Combination With the CDK4/6 Inhibitor Ribociclib, With the PI3K Inhibitor Alpelisib, With the mTOR Inhibitor Everolimus, or With CDK4 Inhibitor Atirmociclib in Adult Subjects With Advanced and/or Metastatic ER Positive, HER2 Negative Breast Cancer
Brief Title: Phase 1b Study of OP-1250 (Palazestrant) in Combination With Ribociclib, Alpelisib, Everolimus, or Atirmociclib in ER+, HER2- Breast Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Olema Pharmaceuticals, Inc. (Industry)
Collaborators: Novartis (Industry); Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OP-1250-003
Record Dates: First submitted 2022-08-16; First posted 2022-08-19 (Actual); Last update posted 2025-10-22 (Actual); Status verified 2025-10

CONDITIONS: Metastatic Breast Cancer; ER-positive Breast Cancer; HER2-negative Breast Cancer; Breast Cancer; Locally Advanced Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — ribociclib; Alpelisib; Everolimus; Sirolimus

STUDY DESIGN:
Intervention Model Description: Treatment Group 1: Palazestrant in combination with ribociclib
  Treatment Group 2: Palazestrant in combination with alpelisib
  Treatment Group 3: Palazestrant in combination with everolimus
  Treatment Group 4: Palazestrant in combination with atirmociclib
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Palazestrant with Ribociclib (Experimental): Treatment Group 1: Palazestrant in combination with ribociclib (KISQALI®, Novartis Pharmaceuticals Corporation).
  Interventions: Drug: Palazestrant; Drug: Ribociclib
- Palazestrant with Alpelisib (Experimental): Treatment Group 2: Palazestrant in combination with alpelisib (PIQRAY®, Novartis Pharmaceuticals Corporation)
  Interventions: Drug: Palazestrant; Drug: Alpelisib
- Palazestrant with Everolimus (Experimental): Treatment Group 3: Palazestrant in combination with everolimus
  Interventions: Drug: Palazestrant; Drug: Everolimus
- Palazestrant with Atirmociclib (Experimental): Treatment Group 4: Palazestrant in combination with atirmociclib
  Interventions: Drug: Palazestrant; Drug: Atirmociclib

INTERVENTIONS:
Drug: Palazestrant — Complete estrogen receptor antagonist (CERAN)
Drug: Ribociclib — All subjects in Treatment Group 1 will receive palazestrant in combination with ribociclib.
  Other Names: KISQALI®; CDK4/6 inhibitor
  Arms: Palazestrant with Ribociclib
Drug: Alpelisib — All subjects in Treatment Group 2 will receive palazestrant in combination with alpelisib.
  Other Names: PIQRAY®; PI3K Inhibitor
  Arms: Palazestrant with Alpelisib
Drug: Everolimus — All subjects in Treatment Group 3 will receive palazestrant in combination with everolimus.
  Other Names: mTOR inhibitor
  Arms: Palazestrant with Everolimus
Drug: Atirmociclib — All subjects in Treatment Group 4 will receive palazestrant in combination with atirmociclib.
  Other Names: CDK4i
  Arms: Palazestrant with Atirmociclib

SUMMARY:
This is a Phase 1b open-label, 2-part study in 3 treatment groups. The 3 treatment groups are as follows:

Treatment Group 1: Palazestrant (OP-1250) in combination with ribociclib (KISQALI®, Novartis Pharmaceuticals Corporation).

Treatment Group 2: Palazestrant (OP-1250) in combination with alpelisib (PIQRAY®, Novartis Pharmaceuticals Corporation).

Treatment Group 3: Palazestrant (OP-1250) in combination with everolimus.

Treatment Group 4: Palazestrant (OP-1250) in combination with atirmociclib.

DETAILED DESCRIPTION:
Part 1 (Dose Escalation): This part will evaluate the safety and pharmacokinetics of a range of doses of palazestrant administered orally (PO) daily to subjects in combination with 600 mg of ribociclib administered PO daily for 21 consecutive days followed by 7 days off treatment (Treatment Group 1) or with 300 mg or 250 mg of alpelisib administered PO daily (Treatment Group 2) or with everolimus 10 mg administered PO daily (Treatment Group 3) and determine the RP2D (Recommended Phase 2 Dose) for each treatment group. Part 1, for Treatment Group 4, will evaluate the safety and pharmacokinetics of OP-1250 at 60 mg or 90 mg doses administered orally (PO) QD in combination with atirmociclib 300 mg PO twice a day (BID).

Part 2 (Dose Expansion): This part of the study will further evaluate the safety and PK of palazestrant at the RP2D in combination with ribociclib (Treatment Group 1), alpelisib (Treatment Group 2), or everolimus (Treatment Group 3) and provide an exploratory estimate of anti-tumor activity of the combinations. An additional group of palazestrant at an alternate dose level in combination with ribociclib (Treatment Group 1b) will be explored to optimize the RP2D of palazestrant. Part 2, for Treatment Group 4, will further evaluate the safety and pharmacokinetics of atirmociclib and OP-1250 at the recommended dose for expansion.

ELIGIBILITY:
Inclusion Criteria:

* Female or male aged >18 years.
* Willing and able to participate and comply with all study requirements.
* Histologically- or cytologically-confirmed advanced or metastatic Breast Cancer (mBC).
* ER+/HER2- disease, as determined in the most recently obtained archival tumor tissue sample from a metastatic site, using locally accepted criteria by the local pathology report.
* Evaluable disease with one of the following: Measurable disease, ie, at least 1 measurable lesion as per RECIST 1.1 (a lesion at a previously irradiated site may only be counted as a target lesion if there is clear sign of progression since the irradiation) OR patients with predominantly bone disease (with or without other non-measurable lesions) are allowed if it is possible to evaluate on radiological examinations (eg. bone scan, PET/CT, CT, MRI) even if lesions are non-measurable according to RECIST 1.1.
* Life expectancy ≥6 months, as judged by the investigator.
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0 or 1.
* Has received no more than 1 prior hormonal regimen (Treatment Group 1). Has received no more than 2 prior hormonal regimens (Treatment Group 2 and Treatment Group 3) . Has received no more than 2 prior hormonal regimens for metastatic disease in Part 1 (Dose Escalation) and no more than 1 prior hormonal regimes in Part 2 (Dose Expansion) for metastatic disease, regardless of type of endocrine agent (Treatment Group 4) for advanced or metastatic disease. Prior hormonal regimens in combination with CDK4/6 inhibitors are allowed in all treatment groups. For subjects in Treatment Group 4, no prior chemotherapy for metastatic breast cancer is allowed.
* Has received no more than 1 prior chemotherapy (which includes antibody drug conjugates) for locally advanced or metastatic breast cancer.

Exclusion Criteria:

* Prior or concurrent malignancy whose natural history or treatment may interfere with the safety or efficacy assessment of the investigational regimen.
* Clinically significant, uncontrolled heart disease and/or cardiac repolarization abnormality.
* History of cerebral vascular disease within 6 months prior to the first administration of study drug dose.
* History of a pulmonary embolism, or deep venous thrombosis within the last 6 months, or subject has an increased risk of thrombosis as determined by the investigator.
* History of pneumonitis or interstitial lung disease.
* Leptomeningeal disease or spinal cord compression.
* Medical history or ongoing gastrointestinal disorders that could affect absorption of oral therapeutics.
* Known human immunodeficiency virus infection.
* Known clinically significant history of liver disease consistent with Child-Pugh Class B or C, including active viral or other hepatitis (eg, hepatitis B or hepatitis C virus), current alcohol abuse, or cirrhosis.
* History of severe cutaneous reaction, such as Stevens-Johnson syndrome, erythema multiforme, toxic epidermal necrolysis, or drug reaction with eosinophilia and systemic symptoms.
* Active infection or at a high risk of developing a serious infection (e.g. participants with immunodeficiencies, uncontrolled diabetes mellitus, uncontrolled heart disease, poor general health, poor nutritional status).
* Has clinically significant co-morbidities, such as, psychiatric disease, or any other condition that could impact the ability of the subject to participate in this study or otherwise has the potential to confound the study results.
* Have received prior treatment with OP-1250.
* Have received prior treatment with approved or investigational PI3K inhibitor (Treatment Group 2) or mTOR inhibitor (Treatment Group 3).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Estimated)
Dates: Start 2022-08-31 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-01-31 (Estimated)

PRIMARY OUTCOMES:
Dose Limiting Toxicities (DLTs) | The first 28 days of treatment
  To determine the maximum tolerated dose (MTD) and/or recommended Phase 2 dose (RP2D), and/ or recommended dose expansion (RDE) of palazestrant when administered with ribociclib (Treatment Group 1), alpelisib (Treatment Group 2), or everolimus (Treatment Group 3), or atirmociclib (Treatment Group 4). The incidence of DLTs will be assessed in the Dose Escalation part (Part 1) of the study.
Characterize the incidence, nature and severity of treatment emergent adverse events (TEAEs) and serious adverse events (SAEs) of palazestrant when administered with ribociclib, alpelisib, everolimus, or atirmociclib. | Up to 30 days after last dose of study drug(s) treatment
  Characterize the incidence, nature and severity of TEAEs and SAEs of palazestrant when administered with ribociclib (Treatment Group 1), alpelisib (Treatment Group 2), everolimus (Treatment Group 3), or atirmociclib (Treatment Group 4) according to NCI-CTCAE version 5.0.
Pharmacokinetics (PK) of palazestrant when administered with ribociclib (Treatment Group 1) or alpelisib (Treatment Group 2), everolimus (Treatment Group 3), or atirmociclib (Treatment Group 4) . | Every 28 days
  To assess the PK of palazestrant (and potential metabolites) in combination with ribociclib (Treatment Group 1), alpelisib (Treatment Group 2), everolimus (Treatment Group 3), or atirmociclib (Treatment Group 4). Plasma levels of palazestrant will be assessed at predefined intervals to establish PK parameters (including: Cmax, Cmin, Tmax, AUC, and t1⁄2 as data permit) and palazestrant trough concentration at steady state).

SECONDARY OUTCOMES:
Preliminarily assess the anti-tumor activity Overall Response Rate of palazestrant when administered with ribociclib, alpelisib, everolimus, or atirmociclib as assessed by the investigator using RECIST v1.1. | Up to 1 year
  Tumor response will be evaluated in patients with measurable or evaluable disease using RECISTv1.1 guidelines.
Evaluate clinical benefit rate (CBR) of palazestrant when administered with ribociclib (Treatment Group 1), alpelisib (Treatment Group 2), or everolimus (Treatment Group 3), or atirmociclib (Treatment Group 4). | Up to 1 year
  CBR will be assessed as proportion of subjects achieving complete response (CR), partial response (PR), or stable disease (SD) with duration of at least 24 weeks.
Evaluate duration of response (DoR) of palazestrant when administered with ribociclib (Treatment Group 1), alpelisib (Treatment Group 2), everolimus (Treatment Group 3), or atirmociclib (Treatment Group 4). | Up to 1 year
  DoR will be calculated as the number of days from the start date of PR or CR (whichever response is achieved first) to the first date that progressive disease is documented.

CONTACTS AND LOCATIONS:
Overall Officials: Daniela Vecchio, PhD, Study Director — Olema Pharmaceuticals, Inc.
Locations (16):
- United States (14):
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - University of California San Francisco Health, San Francisco, California
  - University of Colorado Cancer Center, Aurora, Colorado
  - Advent Health Hematology and Oncology, Orlando, Florida
  - University of Iowa, Iowa City, Iowa
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Henry Ford Health, Detroit, Michigan
  - Regents of the University of Minnesota, Minneapolis, Minnesota
  - Washington University, School of Medicine, St Louis, Missouri
  - Ichan School of Medicine at Mount Sinai, New York, New York
  - Atrium Health Levine Cancer Institute, Charlotte, North Carolina
  - Henry-Joyce Cancer Clinic, The Vanderbilt Clinic, Nashville, Tennessee
  - MD Anderson Cancer Center, Houston, Texas
  - Northwest Medical Specialties, Tacoma, Washington
- Australia (2):
  - Macquarie Health, Sydney, New South Wales
  - Breast Cancer Research Center- Western Australia, Nedlands, Western Australia

IPD SHARING:
Plan to Share IPD: Undecided